CLINICAL TRIAL: NCT00005640
Title: Lymphatic Mapping and Sentinel Lymph Node Biopsy in the Treatment of Colorectal Cancer: A Feasibility Study
Brief Title: Lymphatic Mapping and Sentinel Lymph Node Biopsy in the Treatment of Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MCC-11785; NCI-G00-1780 (Other: NCI)
Record Dates: First submitted 2000-05-02; First posted 2004-05-26 (Estimated); Last update posted 2012-09-25 (Estimated); Status verified 2012-09

CONDITIONS: Colorectal Cancer
Keywords: stage I colon cancer; stage II colon cancer; stage III colon cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Technetium Tc 99m Sulfur Colloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mapping and Biopsy (Experimental): Lymph node mapping and sentinel lymph node biopsy. Patients undergo preoperative endoscopy with injection of technetium Tc 99m sulfur colloid around tumor followed by celiotomy and intraabdominal exploration. At 30 minutes following injection, patients undergo lymphatic mapping with a gamma probe and biopsy of the sentinel lymph node(s). Following biopsy and mapping, patients undergo resection of primary tumor.
  Interventions: Procedure: Preoperative Endoscopy; Radiation: Technetium Tc 99m Sulfur Colloid; Procedure: Gamma Probe; Procedure: Biopsy of Sentinel Lymph Nodes

INTERVENTIONS:
Procedure: Preoperative Endoscopy
Radiation: Technetium Tc 99m Sulfur Colloid
Procedure: Gamma Probe
Procedure: Biopsy of Sentinel Lymph Nodes

SUMMARY:
RATIONALE: Diagnostic procedures, such as lymph node mapping and biopsy, may improve the ability to detect the extent of colorectal cancer.

PURPOSE: Diagnostic trial to study the feasibility of lymph node mapping and sentinel lymph node biopsy in patients who have stage I, stage II, or stage III colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the feasibility of lymphatic mapping and sentinel lymph node biopsy in patients with stage I, II, or III colorectal cancer. II. Evaluate technetium Tc 99m sulfur colloid as a mapping agent in this patient population. III. Identify patients with histologically negative nodes but have positive nodes on further detailed examination.

OUTLINE: Patients undergo preoperative endoscopy with injection of technetium Tc 99m sulfur colloid around tumor followed by celiotomy and intraabdominal exploration. At 30 minutes following injection, patients undergo lymphatic mapping with a gamma probe and biopsy of the sentinel lymph node(s). Following biopsy and mapping, patients undergo resection of primary tumor. Patients are followed postoperatively, every 4-6 months for 2 years, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Preoperative diagnosis of stage I, II, or III colorectal cancer No more than 90 days since diagnosis No tumor involving adjacent structures (T4 lesion) No clinical or radiological evidence of stage IV disease No total excision of primary tumor at diagnosis

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Not specified Hepatic: No severe decompensated liver disease, including cirrhosis Renal: Not specified Other: No known primary or secondary immunodeficiencies No other medical conditions or evidence of infection that would preclude study Not pregnant Negative pregnancy test

PRIOR CONCURRENT THERAPY: See Disease Characteristics No prior colonic, aortic, or retroperitoneal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 1999-06; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

PRIMARY OUTCOMES:
Number of Procedures Resulting in Improved Detection | 18 months
  Determine the feasibility of lymphatic mapping and sentinel lymph node biopsy in patients with stage I, II, or III colorectal cancer. Evaluate technetium Tc 99m sulfur colloid as a mapping agent in this patient population. Identify patients with histologically negative nodes but have positive nodes on further detailed examination.

CONTACTS AND LOCATIONS:
Overall Officials: Timothy J. Yeatman, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States